CLINICAL TRIAL: NCT03937570
Title: The Effects of Echo-optimization of Left Ventricular Assist Devices on Functional Capacity, a RAndomized Controlled Trial (VAFRACT)
Brief Title: Effects of Echo-optimization of Left Ventricular Assist Devices on Functional Capacity (VAFRACT)
Acronym: VAFRACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universita di Verona (Other)
Responsible Party: Principal Investigator, Marzia Lilliu, MD, Principal Investigator, PhD student in Cardiovascular Sciences, Universita di Verona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1397CESC
Record Dates: First submitted 2019-05-01; First posted 2019-05-03 (Actual); Results first posted 2021-11-02 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Heart Failure
Keywords: left ventricular assist device; echo-optimization; functional capacity; cardiopulmonary exercise test
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- EO GROUP (Experimental): Patients underwent LVAD echo-optimization; the optimal device speed is confirmed at the end of procedure.
  Interventions: Device: echo-optimization
- CONTROL GROUP (No Intervention): Patients underwent LVAD echo-optimization, but the optimal device speed is not confirmed at the end of procedure.

INTERVENTIONS:
Device: echo-optimization — LVAD echo-optimization consists of routine comprehensive transthoracic echocardiography at the baseline speed setting, followed by stepwise incremental adjustments to the LVAD speed (revolutions per minute: rpm), with collection of prespecified echocardiographic parameters at each new speed (eg, left ventricle end-diastolic diameter, interventricular septal position, aortic valve opening frequency/duration, tricuspid and/or mitral regurgitation severity). The optimal velocity is defined as the one that allows an intermittent aortic valve opening and a neutral position of the interventricular septum without increasing aortic or tricuspid regurgitation, associated or not to a dilatation of the right ventricle. The recommended speed range varies according to the indications given in the data sheet for each specific device.
  Arms: EO GROUP

SUMMARY:
After the implantation of a left ventricular assist device (LVAD), many patients continue to experience exercise intolerance. LVAD echo guided optimization (EO) determines a more favorable hemodynamic profile and could provide an improvement on functional capacity (FC). VAFRACT is a prospective randomized trial to evaluate the additional benefit of an EO approach on FC, measured by cardiopulmonary exercise test (CPET), in LVAD optimization free population.

DETAILED DESCRIPTION:
The use of Left Ventricular Assist Devices (LVAD) is a viable therapeutic option to improve survival and quality of life of patients with advanced and refractory heart failure (HF). However, after the implantation of an LVAD, patients' functional capacity (FC) is still reduced with maximum oxygen uptake (VO2 peak) values calculated at the cardiopulmonary exercise test (CPET) ranging from 11 to 20 ml/kg/min. LVAD echo guided optimization (EO) determines a more favorable hemodynamic profile, in particular for the right ventricle, and could provide an improvement on FC. VAFRACT is a prospective randomized trial to evaluate the additional benefit of an EO approach on FC, measured by CPET in LVAD optimization free population.

The optimal device speed is defined as the one that allows an intermittent aortic valve opening and a neutral position of the interventricular septum without increasing aortic or tricuspid regurgitation associated or not to a dilatation of the right ventricle (RV). In this condition it is reasonable to expect a more favorable hemodynamic profile for the RV and a better response in terms of functional capacity.

Subjects studied are HF patients supported with a continuous-flow LVAD: HeartMate II (Thoratec Inc., Pleasanton, CA) and HeartMate 3 (HM 3, Abbott, North Chicago, IL). Patients are recruited from our Day Hospital of the Cardiac Surgery Department at the University Hospital of Verona.

ELIGIBILITY:
Inclusion Criteria:

* at least 3 months after LVAD implantation;
* compliance to the required follow-up schedule;
* age 18 or above or of legal age to give informed consent specific to state and national laws.

Exclusion Criteria:

* distance of less than 150 meters on the six-minute walk test (6MWT) or impossibility to perform CPET
* recent finding of any major device-related complication (sepsis, thrombosis …).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2018-02-08 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MARZIA LILLIU, MD, Principal Investigator
Locations (1):
- Department of Cardiac Surgery, University of Verona, Verona, Italy

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | EO GROUP | CONTROL GROUP
Started | 13 | 14
Completed | 13 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EO GROUP | CONTROL GROUP | Total
Number analyzed (Participants) | 13 | 14 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 3 | 4 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.3 (10) | 63 (6.4) | 61.7 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 12 | 13 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 00 | 0
  White | 13 | 14 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Italy | 13 | 14 | 27
VO2 peak [Mean (Standard Deviation); unit: mL/kg/min] | 13.2 (2.5) | 13.8 (2.4) | 13.5 (2.4)

OUTCOME MEASURES:

1. Primary Outcome: VO2 Peak
Description: peak oxygen uptake measured by cardiopulmonary exercise test
Time Frame: three months
Measure: Mean (Standard Deviation); unit: mL/Kg/min
Arm/Group | EO GROUP | CONTROL GROUP
Number analyzed (Participants) | 13 | 14
mL/Kg/min
  BASELINE | 13.2 (2.5) | 13.8 (2.4)
  3 MONTHS-FOLLOW UP | 14.2 (2.5) | 13.2 (2.6)

2. Secondary Outcome: Number of Participants With LVAD-related Hospitalizations
Description: Rate of hospitalizations for: device thrombosis, hemorrhagic events, infections, right heart failure, arrhythmias.
Time Frame: Three months
Measure: Count of Participants; unit: Participants
Arm/Group | EO GROUP | CONTROL GROUP
Number analyzed (Participants) | 13 | 14
Participants | 0 | 0

3. Secondary Outcome: QoL: The EQ-5D Questionnaire
Description: Changes in quality of life perceived by EuroQoL (quality of life) Scale. It is an instrument which evaluates the quality of life measuring with one question: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The answers given to these question (1 = no problems; 2 = some problems; 3 = extreme problems) are converted into EQ-5D index, an utility scores anchored at 0 for death and 1 for perfect health. The EQ-5D questionnaire also includes a Visual Analog Scale (VAS), by which respondents can report their perceived health status with a grade ranging from 0 (the worst possible health status) to 100 (the best possible health status).
Time Frame: Three months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EO GROUP | CONTROL GROUP
Number analyzed (Participants) | 13 | 14
score on a scale
  BASELINE | 0.796 (0.1) | 0.804 (0.09)
  3 MONTHS-FOLLOW UP | 0.85 (0.08) | 0.8 (0.08)

4. Secondary Outcome: Nt-proBNP
Description: Nt-proBNP levels
Time Frame: Three months
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | EO GROUP | CONTROL GROUP
Number analyzed (Participants) | 13 | 14
ng/L
  BASELINE | 1743 (1453) | 1759 (1154)
  3 MONTHS-FOLLOW UP | 1484 (1251) | 1538 (1020)

5. Secondary Outcome: Right Ventricular Function
Description: Fractional area change of right ventricle assessed by echocardiography
Time Frame: Three months
Measure: Mean (Standard Deviation); unit: percentage of fractional area change
Arm/Group | EO GROUP | CONTROL GROUP
Number analyzed (Participants) | 13 | 14
percentage of fractional area change
  BASELINE | 36.5 (3.8) | 35.8 (4.1)
  3 MONTHS-FOLLOW UP | 36.8 (3.2) | 35.7 (4.2)

6. Secondary Outcome: CPET Exercise Time
Description: Cardiopulmonary exercise time
Time Frame: Three months
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | EO GROUP | CONTROL GROUP
Number analyzed (Participants) | 13 | 14
seconds
  BASELINE | 490 (98) | 504 (103)
  3 MONTHS-FOLLOW UP | 526 (116) | 499 (107)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | EO GROUP | CONTROL GROUP
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/14
Other Adverse Events (participants affected / at risk) | 0/13 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-19): https://cdn.clinicaltrials.gov/large-docs/70/NCT03937570/Prot_SAP_000.pdf